CLINICAL TRIAL: NCT02186054
Title: Enhancement of T2 Weighted Imaging of the Liver With Fast Spin Echo Magnetic Resonance Imaging (MRI).
Brief Title: T2 Weighted Imaging of the Liver With Fast Spin Echo MRI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial Logistics
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: T2 Weighted MRI Liver
Record Dates: First submitted 2014-07-04; First posted 2014-07-10 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Liver Disease
Keywords: Abdominal-Pelvic MRI (magnetic resonance image); T2W (T2 weighted); FSE Flex (recently developed MRI pulse sequence); Enhanced single shot FSE (fast spin echo).
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imaging- MRI examinations (Other): Liver MRI imaging will be performed on 50 patients.
  Interventions: Device: MRI examinations

INTERVENTIONS:
Device: MRI examinations — Consented patients will be required to stay in the MRI scanner to complete the 2 additional sequences once their standard exam is completed.
  Other Names: MRI; FSE Flex; Enhanced single shot FSE (eSSFSE)

SUMMARY:
The purpose of this study is to test two new MRI (magnetic resonance imaging) sequences to see how they compare to previously used imaging sequences as they may improve the quality of abdominal MRI.

DETAILED DESCRIPTION:
* Approximately 50 patients undergoing routine liver MRI in our practice imaged with one of our 4 clinical scanners will undergo our standard liver MRI protocol with the addition of 2 breath-hold sequences (FSE Flex and eSSFSE) only increasing the scan time by approximately 3 minutes.
* Data will be retrieved from examinations that have been performed from the patient's electronic imaging file stored in our picture archiving and communication system (PACS).
* Images will be completely anonymized. No patient identifiers will be available on the images during the analysis.
* Analyses will include the visual assessment of image quality, presence and severity of imaging artifact and other non-invasive imaging outcomes performed by radiologists blinded to patient information and the type of sequence performed. Data will be presented in a Likert type scale (1=poor, 2=suboptimal, 3=average, 4=above average and 5=excellent) and imaging parameters will be compared using the Wilcoxon sign rank test.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing routine liver MRI imaged with one of our 4 clinical scanners (MR 750W, General Electric, Milwaukee WI)

Exclusion Criteria:

* Patients not undergoing routine liver MRI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The number of abdominal MRI scans deemed improved quality | Regular scan time with one of 4 clinical scanners plus 3 additional minutes
  Data is presented in a Likert type scale (1=poor, 2=suboptimal, 3=average, 4=above average and 5=excellent) and imaging parameters are compared using the Wilcoxon sign rank test.

SECONDARY OUTCOMES:
The number of MRI scans that display severity of imaging artifact | Regular scan time with one of 4 clinical scanners plus 3 additional minutes
  Data is presented in a Likert type scale (1=poor, 2=suboptimal, 3=average, 4=above average and 5=excellent) and imaging parameters are compared using the Wilcoxon sign rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Schieda, MD, Principal Investigator — OHRI
Locations (1):
- Ottawa Hospital (Civic Campus), Ottawa, Ontario, Canada